# **Statistical Analysis Plan**

Clinical Trial Protocol Identification No.

MS200084 0009

**Title:** A Randomized, Open-label, 2-way-crossover Study Assessing

the Bioequivalence between Single Doses of 500 mg Glucophage Immediate Release (GIR) Tablets (Sino-American Shanghai Squibb Pharmaceuticals Ltd./ Manufactured in China) and 500 mg GIR Tablets (Merck Santé in Semoy/ Manufactured in France) under Fed and

Fasted State in Two Groups of Healthy Subjects

Trial Phase I

**Investigational Medicinal** 

Product(s)

Glucophage Immediate Release (GIR)

Clinical Trial Protocol

Version

17 November 2017 / Version 2.0

Statistical Analysis Plan

Author

PPD Biostatistician

PPD Biostatistician

PPD Pharmacokineticist

PPD Pharmacokineticist

Statistical Analysis Plan Date and Version 29 January 2018/Version 1.0

Statistical Analysis Plan Reviewers

PPD

, Senior Biostatistician, PPD

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies. It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2017 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

## 1 Signature Page

## Statistical Analysis Plan (29Jan2018, Final Version 1.0): MS200084\_0009

**Shells (29Jan2018, Final Version 1.0):** MS200084 0009

A Randomized, Open-label, 2-way-crossover Study Assessing the Bioequivalence between Single Doses of 500 mg Glucophage Immediate Release (GIR) Tablets (Sino-American Shanghai Squibb Pharmaceuticals Ltd./ Manufactured in China) and 500 mg GIR Tablets (Merck Santé in Semoy/Manufactured in France) under Fed and Fasted State in Two Groups of Healthy Subjects

| PPD : |
|-----------------------------------------------------|
| Trial Biostatistician |
| Merck-Serono (Beijing) Pharmaceutical R&D Co., Ltd. |
| Signature: Date: |
| PPD Trial Biostatistician |
| PPD |
| Signature: Date: |
| Senior Statistical Reviewer |
| PPD |
| Signature: Date: |
| CRO Pharmacokineticist |
| PPD |
| Signature: Date: |

| PP | D |
|----|---|

CRO Biostatistician

PPD

Signature: Date:

| 2 | Table of Contents | |
|--------|--------------------------------------------------------------|------|
| 1 | Signature Page | 2 |
| 2 | Table of Contents | 4 |
| 3 | List of Abbreviations and Definition of Terms | 6 |
| 4 | Modification History | 9 |
| 5 | Purpose of the Statistical Analysis Plan | 9 |
| 6 | Summary of Clinical Trial Features | 9 |
| 7 | Sample Size/Randomization | 12 |
| 7.1 | Sample Size | 12 |
| 7.2 | Randomization | 14 |
| 8 | Overview of Planned Analyses | 14 |
| 9 | Changes to the Planned Analyses in the Clinical Trial Protoc | ol14 |
| 10 | Protocol Deviations and Analysis Sets | 15 |
| 10.1 | Definition of Protocol Deviations | 15 |
| 10.2 | Definition of Analysis Sets and Subgroups | 15 |
| 11 | General Specifications for Statistical Analyses | 16 |
| 12 | Trial Subjects | 21 |
| 12.1 | Disposition of Subjects and Discontinuations | 21 |
| 12.2 | Protocol Deviations | 21 |
| 12.2.1 | Important Protocol Deviations | 21 |
| 13 | Demographics and Other Baseline Characteristics | 22 |
| 13.1 | Demographics | 22 |
| 13.2 | Medical History | 22 |
| 13.3 | Other Baseline Characteristics | 23 |
| 14 | Previous or Concomitant Medications/Procedures | 23 |
| 15 | Treatment Compliance and Exposure | 23 |
| 16 | Endpoint Evaluation | 24 |
| 16.1 | Primary Endpoint Analyses | 24 |
| 16.2 | Secondary Endpoint Analyses | 25 |
| 16.3 | Other Endpoint Analyses | 25 |
| 16.3.1 | Analysis of PK Endpoints | 25 |

# GIR/China & GIR/France MS200084\_0009

| 16.3.2 | Estimation of Individual Pharmacokinetic Parameters by Noncompartmental Analysis | 26 |
|---|---|---|
| 16.3.3 | Analysis of PD Endpoints and Biomarker | 28 |
| 16.3.4 | PK/PD Modelling and Simulation | 29 |
| 16.3.5 | Analysis of Molecular Marker | 29 |
| 17 | Safety Evaluation | 29 |
| 17.1 | Adverse Events | 29 |
| 17.1.1 | All Adverse Events | 30 |
| 17.1.2 | Adverse Events Leading to Treatment Discontinuation | 30 |
| 17.2 | Deaths, Other Serious Adverse Events, and Other Significant<br>Adverse Events | 31 |
| 17.2.1 | Deaths | 31 |
| 17.2.2 | Serious Adverse Events | 31 |
| 17.3 | Clinical Laboratory Evaluation | 31 |
| 17.4 | Vital Signs | 32 |
| 17.5 | Other Safety or Tolerability Evaluations | 33 |
| 17.5.1 | ECG Evaluation | 33 |
| 17.5.2 | Physical Examinations, and Chest X-ray | 33 |
| 18 | References | 34 |

# 3 List of Abbreviations and Definition of Terms

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| AUC | Area under the plasma concentration-time curve |
| $AUC_{0\to\infty}$ | The AUC from time zero (dosing time) extrapolated to infinity |
| $AUC_{0 o t}$ | The AUC from time zero (= dosing time) to the last sampling time ( $t_{last}$ ) at which the concentration is at or above the lower limit of quantification |
| AUCextra% | The AUC from time $t_{last}$ extrapolated to infinity given as percentage of $AUC_{0\to\infty}$ |
| BE | Bioequivalence |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| $\mathrm{CL}_{/\mathrm{f}}$ | The apparent total body clearance of drug following extravascular administration. |
| $C_{max}$ | Maximum observed plasma concentration |
| CRO | Contract Research Organization |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Report |
| CTMS | Clinical Trial Management System |
| CTP | Clinical Trial Protocol |
| CV | Coefficient of Variation (%) |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| GCP | Good Clinical Practice |
| GeoCV% | Geometric Coefficient of Variation |
| GeoMean | Geometric Mean |
| GIR | Glucophage Immediate Release |
| HR | Hazard ratio |
| HAV | Hepatitis A Virus |
| $HbA_{1C}$ | Glycosylated Hemoglobin Type A <sub>1C</sub> |

HBsAg Hepatitis B Surface Antigen

HCV Hepatitis C Virus

HIV Human Immunodeficiency Virus

ICF Informed Consent Form

ICH International Conference on Harmonization

IMP Investigational Medicinal Product

LLOQ Lower Level of Quantification

Max Maximum

Mean Arithmetic mean

Min Minimum

MedDRA Medical Dictionary For Regulatory Activities

MRI Magnetic Resonance Imaging
MSS Merck Santé s.a.s. in Semoy

N Number of non-missing observations

PK Pharmacokinetics
PR Partial Response
PT Preferred team

SAE Serious Adverse Event

SASS Sino-American Shanghai Squibb Pharmaceuticals Ltd

SAP Statistical Analysis Plan SBP Systolic Blood Pressure

SD Standard Deviation

SDTM Study Data Tabulation Model
SEM Standard Error of the Mean

SOC System Organ Class

t<sub>1/2</sub> Apparent terminal half-lifeT2DM Type 2 Diabetes Mellitus

TEAE Treatment-Emergent Adverse Event

t<sub>last</sub> The last sampling time at which the concentration is at or above

the lower limit of quantification

t<sub>max</sub> The time to reach the maximum observed concentration

TP Treponema Pallidum

| | Apparent volume of distribution during the terminal phase following extravascular administration |
|---|---|
| $\lambda_{\mathrm{z}}$ | Terminal elimination rate constant |

## 4 Modification History

| Unique<br>Identifier for<br>SAP Version | Date of Author SAP Version | | Changes from the Previous Version |
|---|---|---|---|
| Draft V0.1 | 17 November 2017 | PPD | Not Applicable –First Version |
| Draft V0.2 | 01 December 2017 | PPD | Updated based on SBR comments |
| Draft V0.3 | 20 December 2017 | PPD | Updated based on Sponsor comments |
| Draft V0.4 | 12 January 2018 | PPD | Updated based on Sponsor comments |
| Draft V0.5 | 15 January 2018 | PPD | Updated based on Sponsor comments |
| Draft V0.6 | 22 January 2018 | PPD | Updated based on Sponsor comments |

## 5 Purpose of the Statistical Analysis Plan

The purpose of this Statistical Analysis Plan (SAP) is to document technical and detailed specifications for the final analysis of data collected for protocol MS200084\_0009, version 2.0. Results of the analyses described in this SAP will be included in the Clinical Study Report (CSR). Additionally, the planned analyses identified in this SAP will be included in regulatory submissions or future manuscripts. Any post-hoc, or unplanned analyses performed to provide results for inclusion in the CSR but not identified in this prospective SAP will be clearly identified in the CSR.

The SAP is based upon Section 8 (Statistics) of the trial protocol and protocol amendments and is prepared in compliance with ICH E9.

# **6** Summary of Clinical Trial Features

| Trial Objectives | Primary Objective: |
|---|---|
| | <ul> <li>To assess bioequivalence (BE) between the GIR formulation manufactured in China (test investigational medicinal production [IMP]) and that manufactured in France (reference IM following single oral dose administrations under fasting and the conditions.</li> </ul> |
| | Secondary Objectives: |
| | • To compare additional pharmacokinetic (PK) parameters of GIR after single dose administrations of test and reference products. |
| | To examine the safety and tolerability of GIR after single dose administrations of test and reference products. |

#### **Trial Endpoints**

## **Primary Endpoints:**

 Primary Endpoints will be the PK parameters area under the (plasma) concentration-time curve from time 0 (dosing time) to the last sampling time (t<sub>last</sub>) at which the concentration is at or above the lower limit of quantification (LLOQ) (AUC<sub>0→t</sub>) and maximum plasma concentration observed (C<sub>max</sub>) of metformin, the active ingredient of GIR tablet.

#### **Secondary Endpoints:**

- Pharmacokinetic endpoints: include time of maximum plasma concentration observed ( $t_{max}$ ), half-life ( $t_{1/2}$ ), area under the plasma concentration curve from time 0 to infinity ( $AUC_{0\rightarrow\infty}$ ), the extrapolated part of area under the plasma concentration-time curve ( $AUC_{extra\%}$ ), terminal elimination rate constant ( $\lambda_z$ ), total clearance following extravascular administration (CL/f), and apparent volume of distribution during the terminal phase following extravascular administration ( $V_{z/f}$ ) for metformin, as well as safety and tolerability.
- <u>Safety Endpoints</u>: include adverse events, vital signs (blood pressure, pulse rate, temperature and respiration), laboratory tests (biochemistry, hematology, and urinalysis), electrocardiogram (ECG), physical examination, and concomitant medications.

| Trial Design | This trial is designed as a Phase I, open-label, randomized, 2-period, 2-sequence, crossover trial to assess BE between single oral doses of GIR from different manufacturing facilities, each given concomitantly as a single dose in fasting or fed state. Subjects will be randomized to receive, in each period, either: |
|---|---|
| | <ul> <li>1 tablet of 500 mg GIR (manufactured in Sino-American Shanghai Squibb Pharmaceuticals Ltd. [SASS]/China) or</li> <li>1 tablet of 500 mg GIR (manufactured in Merck Santé in Semoy [MSS]/ France).</li> <li>Drug administration will be done with or without food depending on group allocation to either fed or fasted condition.</li> </ul> |
| | The trial has a duration of approximately 4 weeks including: |
| | <ul> <li>A screening period within 2 weeks before the first GIR administration</li> <li>First dosing/sampling period up to 2 days (48 hours) after dosing</li> <li>A wash-out period of approximately 7 days after the first GIR administration</li> <li>Second dosing/sampling period up to 2 days (48 hours) after</li> </ul> |
| | dosing A conditional follow-up examination period (only for subjects who has AE during the trial and ongoing at discharge) up to 7 days following the last IMP administration. |
| Planned number of subjects | A total of 44 healthy male and female Chinese subjects will be enrolled in the trial, with each gender representing no less than 1/4 of the total number (also evenly allocated to fasting vs. fed group), and are statistically powered to provide adequate sample size for BE testing. |
| Treatment and Trial Duration | The trial has a duration for each subject of approximately 4 weeks, including: |
| | • A screening period within 2 weeks before the first IMP administration |
| | • First dosing/sampling period up to 2 days (48 hours) after dosing |
| | • A washout period of at least 7 days after the first IMP administration |
| | <ul> <li>Second dosing/sampling period up to 2 days (48 hours) after dosing</li> </ul> |
| | • A conditional follow-up examination period (only for subjects who has AE during the trial and ongoing at discharge) up to 7 days following the last IMP administration. |

| | 14 days prior to the first IMP administration on Day 1) followed by 2 |
|---|---|
| Pharmacokinetics | The plasma concentrations of metformin will be determined by a |
| | validated LC/MS analytical method. Pharmacokinetic parameters |
| | (Primary and Secondary Endpoints) will be calculated according to |
| | non-compartmental analysis methods. The mixed trapezoidal rule will be |
| | used to calculate the area under the plasma concentration curve. |
| Randomization | A total of 44 eligible healthy male and female Chinese subjects (26 in |
| and Blinding | fasting state and 18 in fed state) who meet the eligibility criteria will be |
| and Dimunig | randomized (with each gender representing no less than 1/4 of the total number within each group) on Day 1, in a 1:1 ratio to 1 of 2 treatment sequences: Sequence A-B or Sequence B-A. |
| | As this is an open-label trial, no method of blinding was used. |

## 7 Sample Size/Randomization

## 7.1 Sample Size

The BE is declared if all comparisons in primary hypothesis achieve the criteria - the 90% confidence intervals (CI) for the ratios between test and reference of geometric means of both  $AUC_{0\rightarrow t}$  and  $C_{max}$  for metformin in plasma are within 80.00% to 125.00% in both the fasted and fed group.

Based on the results of previously conducted BE trial PK data, (Iran BE 2013 [fasted] and EML056023-H105 [fed]) [1,2], Glucophage/metformin IR formulation has shown relatively low intra-individual Coefficient of Variation (CV), as shown below (Table and Table).

#### **IRAN BE-2013**

- Test: Single dose of metformin IR 500 mg tablets manufactured by PPD (Iran) under fast condition
- Reference: Single dose of metformin IR 500 mg tablets manufactured by Merck (Darmstadt) under fast condition

Table 1 Results from IRAN Bioequivalence Study-2013 Fasting (n= 21)

| Parameter | Intra-Subject CV<br>(%) | Geometric Mean | | – Ratio <sup>a</sup> (%) | 90% Confidence Limits <sup>a</sup> (%) | |
|---|---|---|---|---|---|---|
| | | Test | Reference | - Natio (70) | Lower | Upper |
| C <sub>max</sub> | 17.5 | 1404.5 | 1425.5 | 102 | 92.14 | 110.95 |
| $AUC_{0 \rightarrow t}$ | 13.8 | 7946.5 | 8049.5 | 100 | 92.72 | 107.37 |

 $AUC_{0\rightarrow t}$  = area under the plasma concentration-time curve from time 0 to time t;  $C_{max}$ = the maximum plasma concentration observed; CV= Coefficient of Variation

<sup>&</sup>lt;sup>a</sup> Results from ANOVA Model



As shown in Table and Table , if applying these CVs together with applicable BE criteria for  $AUC_{0\rightarrow t}$  and  $C_{max}$  [0.80 – 1.25], and CCI

In total, 44 subjects should be included in the trial.

Table 3 Sample size and power – Assuming Coefficient of Variation = 17.5% for  $C_{max}$  and 13.8% for  $AUC_{0\rightarrow t}$  (Iran BE 2013 Fasting) and assume 5% variation for all ratios (95% to 105%)

| Fasted Condition | | | |
|---|---|---|---|
| Power (%) | | | |
| Sample Size | C <sub>max</sub> | $AUC_{0 \rightarrow t}$ | Joint Power |
| 18 | 88.2 | 97.4 | > 85.9 |
| 20 | 91.3 | 98.4 | > 89.9 |
| 22 | 93.6 | 99.0 | > 92.7 |

 $\mathrm{AUC}_{0\rightarrow t}$  = area under the plasma concentration-time curve from time 0 to time t;  $C_{max}$ = the maximum plasma concentration observed



## 7.2 Randomization

Each eligible subject will be allocated to a treatment sequence according to a computer-generated randomization schedule. Subjects will be identified only by their assigned subject number. The subjects will receive consecutive subject numbers in the order of their enrollment into the trial.

A total of 44 eligible healthy male and female Chinese subjects (26 in fasting state and 18 in fed state, Table ) who meet the eligibility criteria will be randomized (with each gender representing no less than 1/4 of the total number within each group) on Day 1, in a 1:1 ratio to 1 of 2 treatment sequences: Sequence A-B or Sequence B-A as presented in Table .

In sequence A-B, subjects will receive test GIR tablets (Treatment A) in Period 1 and reference GIR tablets (Treatment B) in Period 2. In sequence B-A, subjects will receive reference GIR tablets in Period 1 and test GIR tablets in Period 2 after Washout.

**Table 5** Randomization Allocation

| | Day 1 of Period 1 | Day 1 of Period 2 |
|-----------------------|---------------------|---------------------|
| Easting grown (n= 26) | Treatment A (n= 13) | Treatment B (n= 13) |
| Fasting group (n= 26) | Treatment B (n= 13) | Treatment A (n= 13) |
| F. J (n = 10) | Treatment A (n= 9) | Treatment B (n= 9) |
| Fed group (n= 18) | Treatment B (n=9) | Treatment A (n=9) |

Subjects will only be replaced if the number of subjects within each group falls below 20 (fasting) or 12 (fed). The subject who is replacing a discontinued subject will then be allocated to the treatment sequence of the subject who discontinued.

# 8 Overview of Planned Analyses

The methods described in this document will be applied to the preparation of tables, figures and listings (TLFs). Statistical analyses will be performed using cleaned electronic clinical report form (eCRF) data collected.

This SAP will cover the final analysis only. The final analysis will be performed only after the last subject has completed the study with all study data in-house and all data queries resolved. The SAP will be finalized prior to database lock.

# 9 Changes to the Planned Analyses in the Clinical Trial Protocol

The Screening Population has been added to include all subjects who signed informed consent in the study.

## 10 Protocol Deviations and Analysis Sets

#### 10.1 Definition of Protocol Deviations

Protocol deviations describe how close the study has been conducted according to the protocol as expected per GCP. Some of these deviations may be significant contributors to analysis bias.

Important protocol deviations are protocol deviations that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a subject's rights, safety, or well-being.

Examples of clinically important protocol deviations or important events for PK include, but may not be limited to, the following:

- Subjects that are dosed on the study despite not satisfying the inclusion criteria
- Subjects that develop withdrawal criteria whilst on the study but are not withdrawn
- Subjects that receive the wrong treatment or an incorrect dose
- Subjects that receive an excluded concomitant medication
- Vomiting following oral dosing (handling of this event is described under Section 10.2; each instance will be discussed in the CSR)
- Deviation from GCP
- Sample processing errors that may lead to inaccurate bioanalytical results
- Failure to fast (in fasted arm) or incomplete meal consumption (in fed arm) prior to dosing

The following deviations will be identified and confirmed prior to or at the Data Review Meeting at the latest. Important protocol deviations include:

- Deviations from the inclusion and exclusion criteria
- Deviations post inclusion

A data review meeting will be held to discuss and update the definition of important protocol deviations so as to determine the evaluability of the subjects prior to database lock.

# 10.2 Definition of Analysis Sets and Subgroups

#### **Screening Population**

The Screening population includes all subjects who have signed the main informed consent (i.e., screening failures plus subjects enrolled).

#### **Safety Population**

The Safety Population includes all subjects who received at least 1 dose of IMP. In general, clinical data will be analyzed for the Safety Population.

#### **Pharmacokinetic Population**

The PK Analysis Set includes all subjects who completed the trial with adequate trial medication compliance, without any relevant protocol violations or events with respect to factors likely to affect the comparability of PK results, and with sufficient evaluable data to determine primary endpoints (AUC<sub>0 $\rightarrow$ t</sub> and C<sub>max</sub>) for both treatments. If subjects receive concomitant medication that potentially affects PK for the treatment of an AE, their inclusion in the PK Analysis Set will be decided on a case-by-case basis. Emesis occurring within two times of the median t<sub>max</sub> for a given treatment will be considered a relevant event likely to affect the comparability of PK results. Similarly, a predose concentration for a given treatment period which exceeds 5% of C<sub>max</sub> will be considered a relevant event affecting PK results. All PK analyses will be based on the PK Analysis Set. Data for subjects excluded from the PK Analysis set will be included in listings.

## 11 General Specifications for Statistical Analyses

#### **Output Presentations:**

The shells provided with this SAP describe presentations for this study and therefore the format and content of the summary tables, listings and figures to be provided by IQVIA Biostatistics. Unless otherwise indicated all analyses will be presented separately for the two treatments (Treatment A and Treatment B) and for two treatment sequences (Sequence A-B and Sequence B-A) under different food condition (fed and fasted).

#### Listings

All listings will be reported separately by food condition and sorted by treatment or treatment sequence (A-B or B-A), and/or scheduled time point, as appropriate. Data which are only collected before administration of trial drug and/or at end of study will be sorted by subject and scheduled time point (if appropriate).

All PK concentrations will be reported and analyzed with the same precision as the source data provided by the bioanalytical laboratory or clinical laboratory regardless of how many significant figures or decimal places the data carry. In export datasets, as well as in the Study Data Tabulation Model (SDTM) PP/XD domain, PK parameters will be provided with full precision, and will not be rounded.

Pharmacokinetic parameters and actual elapsed sample collection times will be rounded for reporting purposes in by-subject listings. Actual elapsed sample collection times will be rounded to two decimal places with units of hours. For PK parameters, the standard rounding procedure will be as follows:

- Parameters directly derived from source data (e.g., C<sub>max</sub>) will be reported and analysed with the same precision as the source data.
- Parameters derived from actual elapsed sample collection times (e.g.,  $t_{max}$ ) will be reported to two decimal places with units of hours.

- Values of AUC will be rounded to 3 significant figures.
- Percentages not derived directly from source data (e.g., AUC<sub>extra</sub>%) will be reported to 3 significant figures.
- Other parameters (e.g.,  $t_{1/2}$ ,  $\lambda_Z$ ,  $CL_{f}$ ,  $V_{z/f}$ ) will be reported with 3 significant figures.

## **Tables and Descriptive Statistics**

All data will be summarized by food condition, treatment or treatment sequence, and/or scheduled time point, as appropriate. Repeated and unscheduled measurements included in the listings will not be used for statistical analyses or summaries, unless the repeated measurement was performed due to unreliable values/technical reasons, e.g., clotted samples. Unscheduled measurements will not be included in by-visit table summaries and graphs, but will contribute to the baseline value and best/ worst case value where required.

Metformin concentration in plasma and its PK parameters will be presented in tables and descriptively summarized by food condition, treatment, and/or nominal time point, as appropriate.

#### **Presentation of PK Concentration Data**

Pharmacokinetic concentration data will be descriptively summarized using: number of non-missing observations (N), arithmetic mean (Mean), standard deviation (SD), standard error of the mean (SEM), CV%, minimum (Min), median (Median) and maximum (Max).

Descriptive statistics of PK concentration data will be calculated using values with the same precision as the source data, and rounded for reporting purposes only. The following conventions will be applied when reporting descriptive statistics of PK concentration data:

Mean, Min, Median, Max:

SD:

4 significant digits

CV%:

1 decimal place

Descriptive statistics of plasma concentrations below the LLOQ will be taken as zero.

#### Presentation of PK Parameter Data

Pharmacokinetic parameter data will be descriptively summarized using: N, Mean, SD, CV%, Min, Median, Max, geometric mean (GeoMean), the geometric coefficient of variation (GeoCV%), and the 95% CI for the GeoMean (LCI 95% GM, UCI 95% GM).

Descriptive statistics of PK parameter data will be calculated using full precision values, and rounded for reporting purposes only.

The following conventions will be applied when reporting descriptive statistics of PK parameter data:

Mean, Min, Median, Max, GeoMean, 95% CI: 3 significant digits

| GeoMean ratio: | 2 decimal places |
|----------------|----------------------|
| SD: | 4 significant digits |
| CV%, GeoCV%: | 1 decimal place |

#### Presentation of continuous and qualitative variables

Continuous variables will be summarized using the following descriptive statistics unless otherwise specified, i.e.,

- Number of subjects (N), number of subjects with non-missing values
- Mean, SD
- Median
- Minimum and maximum

Qualitative variables will be summarized by counts and percentages.

Unless otherwise stated, the calculation of proportions will be based on the number of subjects of the analysis set of interest. Therefore, counts of missing observations will be included in the denominator and presented as a separate category.

In case the analysis refers only to certain visits, percentages will be based on the number of subjects still present in the trial at that visit, unless otherwise specified.

#### **Software:**



All other statistical analyses will be conducted using SAS® Version 9.4 or higher.

#### **Definition of baseline:**

Unless otherwise specified, baseline for end of study is defined as the last non-missing measurement taken prior to or on the day of the first IMP administration (including unscheduled assessments as applicable).

For vital signs, the assessment performed within 4 hours prior to IMP administration in each treatment period will be considered as baseline for the treatment period. If there is no time point, the last non-missing assessment prior to dosing in each period will be taken as baseline.

In the case where the last non-missing measurement and the dosing date/time coincide, that measurement will be considered baseline, but medications commencing on the first IMP administration date will be considered post-baseline.

## **Definition of End of Study**

Unless otherwise specified, end of study is defined as the last measurement taken prior to or on the day of discharge (D10 or any special day for Premature Withdrawal Visit).

#### **Definition of duration:**

Duration will be calculated by the difference of start and stop date + 1 (e.g. survival time (days) = date of death – date of randomization + 1) (if not otherwise specified).

#### **Conversion factors:**

The following conversion factors will be used to convert days into months or years:

1 month = 30.4375 days

1 year = 365.25 days.

#### **Common calculations:**

For quantitative measurements, change from baseline will be calculated as:

Test Value at Visit X – Baseline Value

#### Handling of discontinued subjects and missing data:

Unless otherwise specified, data from discontinued subjects will not be replaced. Handling of missing data for PK parameter calculations are discussed under Section 16.3.2.

In all subject data listings, imputed values will be presented. In all listings imputed information will be flagged.

Missing statistics, e.g. when they cannot be calculated, should be presented as "nd". For example, if n=1, the measure of variability (SD) cannot be computed and should be presented as "nd". If n=2, summaries will not be computed and will be presented as "nd".

For the derivation of new date variables the following rules will apply:

Partial birth dates will be handled this way: day will be imputed as 15 if it is missing, and month imputed as June if missing. If both of day and month are missing, they will be imputed as July 1st. If year is missing then the date will not be imputed.

Any adverse event (AE) with incomplete start/time and or end dates will be handled as described below for the classification as treatment-emergent, assignment to treatment periods, and calculation of duration.

- AE with unknown start time but known start date, will be imputed with a time of 00:00 hours, unless the start date corresponds to any given dosing date, in which case time of dosing will be used instead. However, if this results in a start time after end time of the AE, then the start time will be imputed to 00:00 hours instead.
- Any AE with completely unknown start date will be imputed with date and time of the first IMP administration, unless the end date (imputed if needed) is known and prior to first IMP administration. In the latter case, the start date will be missing.
- AE with partially missing start date but in the same year (when day and month are missing) or in the same month and year (if the day is missing) as first IMP administration then the start date will be replaced by the minimum between first IMP administration and AE resolution date. In all other cases the missing onset day or onset month will be replaced by 01.
- Adverse event with completely unknown end date will be imputed with the date of study completion (or in case of withdrawal, date of discontinuation).

Partially known end dates will be treated as follows:

- If only the day is missing, the last day of the month will be imputed or the date of study completion/discontinuation if earlier.
- If day and month are both missing, then the end date of 31 December will be imputed or the date of study completion/discontinuation if earlier.

Assignment to the different treatment periods will be performed after the imputations have been performed. An AE will be assigned to a specific treatment period if it occurs on or after the IMP administration scheduled for that period and before the IMP administration in the next period (or study completion for the last period).

#### Trial day:

Trial day will be calculated from the reference start date, and will be used to show start/end day of assessments and events. Reference start date is defined as the day of the first IMP administration in period 1. Trial Day 1 is the day of first IMP administration in period 1. The day before is defined as Trial Day -1 (no Trial Day 0 is defined). Trial day will be calculated accordingly:

• If the date of the event is on or after the reference start date then:

Trial day = (date of event - reference start date) + 1.

• If the date of the event is prior to the reference start date then:

Trial day = (date of event - reference start date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, and Trial Day and any corresponding durations will be presented as missing. Rules of handling missing dates relevant to efficacy will specified in the subsequent sections.

## 12 Trial Subjects

This section includes specifications for reporting subject disposition and treatment/trial discontinuations. Additionally, procedures for reporting protocol deviations are provided.

## 12.1 Disposition of Subjects and Discontinuations

All subjects who provide informed consent will be accounted into this study. Subject disposition and withdrawals will be presented for the Screening Population.

The following summaries will be produced by treatment sequence and overall, for each food condition group:

- Total number of subjects screened (i.e. subjects who gave informed consent)
- Numbers of randomized subjects
- Number of subjects treated in each period
- Number of subjects who complete the trial
- Number of subjects who discontinued the study treatment after the first administration, grouped by the main reason
- Number of subjects who terminated the study prematurely, grouped by the main reason
- Number of subjects included in Safety Population
- Number of subjects included in PK Population

Corresponding individual listings will be prepared (sorted by group, treatment sequence and subject).

Additionally, a listing of the screening failures will be produced with the reason of non-inclusion in the treatment phase.

Listings with visit dates will also be carried out by group, treatment sequence and subject.

#### 12.2 Protocol Deviations

# 12.2.1 Important Protocol Deviations

Important protocol deviations will be based on the Clinical Trial Management System (CTMS) data and determined by medical review process. All important protocol deviations will be included in SDTM datasets, if identified through medical review. The Analysis Data Model (ADaM) datasets will be derived from SDTM and include all important protocol deviations.

A data review meeting will be held to discuss and update the definition of important protocol deviations so as to determine the evaluability of the subjects prior to database lock.

The following outputs will be provided by treatment sequence and overall, for each food condition group:

- Summary of important protocol deviations relating to inclusion/exclusion criteria
- Summary of other important protocol deviations post inclusion criteria

All important protocol deviations will be listed. A listing presenting protocol deviations relating to inclusion/exclusion criteria and a listing presenting other deviations will be produced.

## 13 Demographics and Other Baseline Characteristics

Unless otherwise specified, demographic data and other baseline characteristics will be presented for the Safety Population.

Summaries of the key demographics overall and by treatment sequence for each group are to be provided. Continuous variables will be summarized using the descriptive statistics. Qualitative variables will be summarized by counts and percentages. No statistical testing will be carried out for demographic or other baseline characteristics.

## 13.1 Demographics

Demographic characteristics will be summarized using the following information from the Screening/Baseline Visit eCRF pages.

Demographic characteristics

- Age (years): summary statistics
- Sex: Male, Female
- Race: Chinese, Non-Chinese
- Weight (kg): summary statistics
- Height (cm): summary statistics
- BMI (kg/m<sup>2</sup>): summary statistics

Specifications for computation:

- Age (years):
- (date of given informed consent date of birth + 1) / 365.25

# 13.2 Medical History

The medical history will be summarized from the "Medical History" eCRF page, using MedDRA, Version 20.1 or higher version, preferred term (PT) as event category and MedDRA system organ class (SOC) body term as Body System category.

Medical history will be displayed in terms of frequency tables: ordered by primary SOC and PT in alphabetical order.

#### 13.3 Other Baseline Characteristics

The following baseline characteristics will be reported overall and by treatment sequence for each group:

- Nicotine and Alcohol Consumption
- Urine Testing of drugs of abuse
- Breath test of alcohol
- Serology: HAV antibody, HBsAg, HCV antibody, HIV antibody, TP antibody

Baseline characteristics with respect to vital signs, ECG recordings and laboratory tests will be part of Section 17 (Safety Evaluation).

Results of chest x-ray and serum pregnancy test (for women of childbearing potential) will be presented only in the listings.

#### 14 Previous or Concomitant Medications/Procedures

Previous and concomitant medication/ procedure will be tabulated for Safety Population. All medications and procedures will be presented in the listings.

Medications will be coded using World Health Organization Drug Dictionary Enhanced (WHO-DDE) Version 01Sep2017 or higher version. Procedures will be coded using MedDRA Version 20.1 or higher version.

**Previous medications** are medications started and ended before first IMP administration.

**Concomitant medications/ procedures** are medications/ procedures, other than trial medications/ procedures, which are taken by subjects any time on-trial (include medications/ procedures which started before the first IMP administration and were ongoing after first IMP administration, or started on or after the first IMP administration day).

Previous and concomitant medications will be summarized overall for both groups as well as overall and by treatment sequence for each group, and by PT and ATC 2nd level, respectively. The listing of previous and concomitant medications/procedures will be generated.

Concomitant procedures will be summarized overall for both groups as well as overall and by treatment sequence for each group, and by reason for procedure and PT, respectively. The listing of previous and concomitant procedures will be generated.

# 15 Treatment Compliance and Exposure

Safety Population will be used to list the IMP administration. IMP administration will be listed by group, treatment sequence and subject with treatment, date and time of administration.

Missing or partial dates or time for IMP administration will not be imputed.

## 16 Endpoint Evaluation

## 16.1 Primary Endpoint Analyses

The primary endpoints are the following PK parameters calculated from metformin plasma concentrations:

AUC<sub>0→t</sub> of metformin

C<sub>max</sub> of metformin

The null and alternative hypotheses are the following:

$$H_0$$
: for  $AUC_{0-t}$   $\mu_T / \mu_C \le 0.8$  or  $\mu_T / \mu_C \ge 1.25$ , for at least 1 primary endpoint for  $C_{\text{max}}$   $\mu_T / \mu_C \le 0.8$  or  $\mu_T / \mu_C \ge 1.25$ 

$$H_1$$
: for  $AUC_{0-t}$   $0.8 < \mu_T/\mu_C < 1.25$ , for both primary endpoints and for both fasting and fed groups

where  $\mu_T$  and  $\mu_C$  are the means of primary endpoints following test IMP and reference IMP (Treatment A and Treatment B), respectively.

The analysis of primary endpoints will be based on PK Population (Section Error! Reference ource not found.)

The primary endpoints, C<sub>max</sub> and AUC<sub>0→t</sub> in fasting and fed group, will be log-transformed and a mixed-effects model will be applied. The model will include fixed effects for sequence, treatment and period and a random effect of subject nested within sequence. Treatment differences on the log scale will be estimated for the parameters together with their 90% CIs. The least squares means together with their 95% CIs by treatment will also be estimated. Point estimates and CIs will be back-transformed to the original scale for presentation, i.e., ratios of geometric means and corresponding 90% CIs for Treatment A/Treatment B, and geometric means and corresponding 95% CIs by treatment, respectively. Intra-subject CV estimated from the model will also be presented. Bioequivalence will be assessed separately in the fed and in the fasted group, and the trial will be considered successful only if BE is established for both primary parameters in both groups. The BE will be considered established if the 90% CIs for the ratios of geometric means between the investigational product and the comparator fall within 80.00% to 125.00% for all these comparisons.

The following example code could be used:

```
proc mixed data=pkparam;
by food param;
class sequence period trt subjid;
model lnest = sequence period trt /ddfm=kr;
```

```
random subjid(sequence);
estimate 'A vs B' trt 1 -1 /alpha=0.1 cl;
lsmeans trt /alpha=0.05 cl;
run;
```

All primary PK endpoints will be descriptively summarized as described in Section Error! eference source not found. Graphs of individual values and geometric mean will be presented for primary PK parameters versus treatment and food condition. Boxplots will also be created for primary PK parameters versus treatment for the fed and the fasted conditions.

## 16.2 Secondary Endpoint Analyses

All secondary PK endpoints will be descriptively summarized as described in Section 11. The secondary PK endpoints are the following parameters in plasma for metformin:

```
t_{max},\,t_{1/2},\,\lambda_{Z},\,AUC_{0\rightarrow\infty},\,AUC_{extra\%},\,CL/_f,\,V_{z/f}.
```

For  $t_{max}$ , the Hodges-Lehmann estimates for the treatment differences and corresponding 90% CIs according to the Tukey method will be calculated.

The mixed-effects model for treatment comparison as described for the primary endpoints will also be applied to  $AUC_{0\to\infty}$ . The ratios of geometric means and corresponding 90% CIs for Treatment A/Treatment B will be estimated separately for fed and fasted treatments. Graphs of individual  $AUC_{0\to\infty}$  values and geometric mean will be presented by treatment and food condition.

## 16.3 Other Endpoint Analyses

# 16.3.1 Analysis of PK Endpoints

Predose samples that occur before the first drug administration will be assigned a time of 0 hours, as if the sample had been taken simultaneously with the study drug administration.

Pharmacokinetic concentrations which are erroneous due to a protocol deviation (as defined in the protocol), documented handling error or analytical error (as documented in the bioanalytical report) may be excluded from the PK analysis if agreed upon prior to performing a statistical analysis. In this case, the rationale for exclusion must be provided in the Clinical Trial Report (CTR). Any other PK concentrations that appear implausible to the Pharmacokineticist/PKPD Data Analyst must not be excluded from the analysis. Any implausible data will be documented in the CTR.

All statistical analyses and descriptive summaries of PK data will be performed on the PK Analysis Set. Pharmacokinetic concentrations will be listed for all subjects by treatment and fed/fasted group; concentrations excluded from the PK analysis will be flagged within the listing.

A listing of PK blood sample collection times by individual, as well as derived sampling time and time deviations, will be provided.

Plasma concentration data will be summarized descriptively for metformin as described in Section 11. Values below the LLOQ will be taken as zero for descriptive statistics of PK concentrations. Missing concentrations (e.g., no sample, insufficient sample volume for analysis, no result, or result not valid) will be reported and displayed generally as "N.R.".

Samples that are collected outside the specified time windows will be included in the PK analysis but excluded from the concentration summary. The PK sampling collection schedule is presented in Table 6 below.

 Table 6
 Pharmacokinetic Sample Collection Schedule

| Trial Day | Period Day | Time of Blood Sample (hour) | Window<br>Allowance<br>(minute) |
|---|---|---|---|
| 1 | 1 - Predose in Period 1 | Baseline blood draw (10 minutes prior to drug administration) | ±2 |
| 1 | 1 – Single dose administration and Washout begins | 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14 | ±2 |
| 2 | 2 | 24, 36 | ±5 |
| 3 | 3 | 48 | ±5 |
| 4 – 7 | | | |
| 8 | 1-Predose in Period 2 | Baseline blood draw (10 minutes prior to drug administration) | ±2 |
| 8 | 1 – Single dose administration and Washout begins | 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 14 | ±2 |
| 9 | 2 | 24, 36 | ±5 |
| 10 | 3 | 48 | ±5 |
| 11-14 | | | |
| End of Trial (Day<br>15)/Premature<br>Withdrawal | | 1-sample | ±30 |

Individual concentration-time profiles showing all subjects by treatment and fed/fasted group (i.e., individual subject overlay plots), and/or showing all treatment groups by subject (i.e., by-subject plots) will be created using the actual time points and the numeric concentration data. Arithmetic mean concentration-time profiles by treatment and fed/fasted group will be provided using scheduled (nominal) time points and the numeric concentration data. All concentration-time plots for PK data will be presented both on a linear and on a semi-logarithmic scale. Mean plots will include SD error bars when plotted on a linear scale.

# 16.3.2 Estimation of Individual Pharmacokinetic Parameters by Noncompartmental Analysis

For the PK analysis, predose sample concentrations that are below the LLOQ or that are missing will be assigned a numerical value of zero for the calculation of AUC. Any anomalous concentration values observed at predose will be identified in the CTR, and if the anomalous

predose concentration value is greater than 5.00% of the  $C_{max}$  in the profile, the profile will be included in the PK analysis, but the concentration data and the corresponding derived PK parameters will be excluded from summaries and inferential statistics as appropriate; handling of the data will be documented in the CTR.

Pharmacokinetic parameters will be calculated using standard noncompartmental methods. Pharmacokinetic parameters will be calculated and listed for all volunteers who provide sufficient concentration-time data. At least 3 valid, postdose concentration points will be required in the PK profile to obtain any PK parameter estimate.

Pharmacokinetic parameters will be calculated using the actual elapsed time since dosing, given with a precision of 14 significant digits. In cases where the actual sampling time is missing, calculations will be performed using the scheduled time. Otherwise, there will be no further imputation of missing data other than for a missing predose concentration as stated above.

For each subject in the PK Analysis Set the following PK parameters will be calculated for metformin, where appropriate:

| Symbol | Definition |
|---|---|
| $AUC_{0 o t}$ | The AUC from time zero (= dosing time) to $t_{last}$ at which the concentration is at or above the LLOQ. Calculated using the mixed log linear trapezoidal rule (linear up, log down). Units: $ng*h/mL$ . |
| $AUC_{0\to\infty}$ | The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at $t_{last}$ , as estimated using the linear regression from $\lambda_z$ determination. $AUC_{0\to\infty}=AUC_{0\to t}+C_{last\ pred}/\lambda_z$ . Units: $ng*h/mL$ . |
| AUC <sub>extra</sub> % | The AUC from time $t_{last}$ extrapolated to infinity given as percentage of $AUC_{0\to\infty}$ . $AUC_{extra\%} = (extrapolated area/AUC_{0\to\infty})*100$ . The predicted $AUC_{0\to\infty}$ should be used. Units: %. |
| CL/f | The apparent total body clearance of drug following extravascular administration, taking into account the fraction of dose absorbed. $CL_{/f} = Dose_{p.o.}/AUC_{0\rightarrow\infty}$ . The predicted $AUC_{0\rightarrow\infty}$ should be used. The dose amount to be used for this calculation is 500 mg. Units: L/h. |
| C <sub>max</sub> | Maximum observed concentration, taken directly from the observed concentration-time profile. Units: ng/mL. |
| t <sub>max</sub> | The time to reach the maximum observed concentration (unless otherwise defined, take the first occurrence in case of multiple/identical $C_{\text{max}}$ values). Units: h. |

| t <sub>1/2</sub> | Apparent terminal half-life. $t_{1/2} = \ln (2)/\lambda_z$ . Units: h. |
|---|---|
| $V_{z/f}$ | The apparent volume of distribution during the terminal phase following extravascular administration, based on the fraction of dose absorbed. $V_{z/f} = Dose/*AUC_{0\to\infty}*\lambda_z$ ) following single dose. Units: L. |
| $\lambda_z$ | Terminal elimination rate constant. Determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve. Units: h <sup>-1</sup> . |

The following PK parameters will be calculated for diagnostic purposes and listed, but will not be summarized:

- The time interval (h) of the log-linear regression ( $\lambda_{z \text{ lower}}$ ,  $\lambda_{z \text{ upper}}$ ) to determine  $\lambda_{z}$ .
- Number of data points  $(N_{\lambda})$  included in the log-linear regression analysis to determine  $\lambda_z$ .
- Goodness-of-fit statistic (Rsq) for calculation of  $\lambda_z$ .

The regression analysis should contain data from at least 3 different time points in the terminal phase consistent with the assessment of a straight line on the log-transformed scale. Phoenix WinNonlin best fit methodology will be used as standard. The last quantifiable concentration should always be included in the regression analysis, while the concentration at t<sub>max</sub> and any concentrations <LLOQ which occur after the last quantifiable data point should not be used.

The Rsq should be  $\geq$ 0.800 and the observation period over which the regression line is estimated should be at least two-fold the resulting  $t_{1/2}$  itself. If these criteria are not met, then the rate constants and all derived parameters (e.g.,  $AUC_{0\to\infty}$ ,  $AUC_{extra\%}$ , CL/f,  $t_{1/2}$ , and  $V_{z/f}$ .) will be included in the parameter outputs and descriptive statistics but will be flagged and discussed appropriately. Any flags should be included in the study specific SDTM.

To ensure a reliable estimate of the extent of exposure in pivotal trials (e.g., BE),  $AUC_{extra\%}$  should be less than or equal to 20.0%. If  $AUC_{extra\%}$  is greater than 20.0%, all parameters derived using  $\lambda_z$  (i.e.,  $\lambda_z$ ,  $t_{1/2}$ ,  $AUC_{0\to\infty}$ ,  $AUC_{extra\%}$ ,  $V_{z/f}$ , and  $CL_{/f}$ ) will not be included in the calculation of descriptive statistics or statistical analyses.

The dose amount for IMP administered is that of the active, free drug substance only, and is synonymous with the measured analyte. No adjustment for the dose amount value of IMP will be applied when 'dose' is used in calculating PK parameters with formulas needing a dose value.

The Phoenix WinNonlin NCA Core Output will be provided in a separate listing.

# 16.3.3 Analysis of PD Endpoints and Biomarker

Not applicable.

## 16.3.4 PK/PD Modelling and Simulation

Not applicable.

## 16.3.5 Analysis of Molecular Marker

Not applicable.

## 17 Safety Evaluation

Population: Safety Population

The subsections in this section include specifications for summarizing safety endpoints that are common across clinical trials such as adverse events, laboratory tests, ECG recordings and vital signs. Safety analyses will be done on the Safety Population. All safety data will be listed in individual subject listings by group, treatment sequence and subject.

All safety variables will be analyzed using descriptive statistics. For the evaluation of safety parameters, the continuous variables will be summarized descriptively by N, mean, median, SD, Q1-Q3, and minimum and maximum values. Categorical variables will be presented in frequency tables with the counts of observations and corresponding percentages.

#### 17.1 Adverse Events

AEs will be coded using the MedDRA Version 20.1 or higher.

An AE will be considered as 'treatment emergent' if it occurred after the first IMP administration of each period or if it was present prior to first IMP administration but exacerbated after the first IMP administration of each period. All other adverse events will be considered 'pre-treatment'.

In the case where it is not possible to define an AE as TEAE or not, the AE will be classified as TEAE as the most conservative approach.

The AE listings will include the following items:

- System organ class
- Preferred term
- Investigator's description
- Whether the event is treatment-emergent
- Trial treatment at onset of event
- Date and time of onset and resolution

- Duration of the event
- Date and time of last administration before AE
- Study Day
- Severity
- Causality relationship to investigational product
- Outcome
- Action taken to investigational product
- Other action
- Seriousness

#### 17.1.1 All Adverse Events

A summary table describing all the TEAEs occurring during the trial will be produced overall and by group as well as by treatment for each group using frequency of events and number and percentage of subjects experiencing these events overall and by SOC and PT.

Group/SOC terms will be sorted by decreasing total frequency. Preferred terms (PT) within each group/SOC term will likewise be sorted by decreasing total frequency.

In addition, all TEAEs will be tabulated by severity and relationship to IMP in the same manner.

Multiple occurrences of the same TEAE in one subject during the same treatment in the trial will be counted as multiple events in the frequency counts for adverse events. If a subject experiences more than one occurrence of the same AE during the same treatment in the trial, the subject will only be counted once for that treatment using the worst severity and the strongest relationship.

In case a subject had events with missing and non-missing severities, the maximum of the non-missing severities will be displayed. In case all the TEAEs of a subject are all with missing severities then Moderate will be used unless there is any evidence that it should be Severe.

# 17.1.2 Adverse Events Leading to Treatment Discontinuation

AEs leading to permanent discontinuation of IMP will be identified as those records with a response of "Drug Withdrawn" to the item "Action taken with study drug" on the "Adverse Events Details" page of the eCRF.

For AEs leading to discontinuation of IMP, summaries of incidence rates (frequencies and percentages) by SOC and PT will be prepared.

All adverse events leading to trial or treatment discontinuation will be listed by group, treatment sequence and subject including SOC, PT and investigators' verbatim.

# 17.2 Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

#### 17.2.1 **Deaths**

AEs leading to Death are those events which are recorded as "Fatal" to the item "Outcome" on the "Adverse Events Details" page of the eCRF. AEs leading to deaths will be listed by group, treatment sequence and subject including SOC, PT and investigators' verbatim, if applicable.

#### 17.2.2 Serious Adverse Events

Serious adverse events (SAEs) are those events recorded as "Yes" to the item "Serious adverse event" on the "Adverse Events Details" page of the eCRF. All SAEs will be listed by group, treatment sequence and subject including SOC, PT and investigators' verbatim.

## 17.3 Clinical Laboratory Evaluation

Results from the central laboratory will be included in the reporting of this study for hematology, biochemistry, and urinalysis. Laboratory evaluations to be included in the outputs are as below:

<u>Hematology</u>: Erythrocytes, Hemoglobin, Hematocrit, Mean corpuscular volume, Mean corpuscular hemoglobin, Mean corpuscular hemoglobin concentration, Red blood cell distribution width, Platelets, Mean platelet volume, Thrombocytocrit, Platelet distribution width, White blood cells, Neutrophils, Monocytes, Lymphocytes.

Biochemistry: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Total Bilirubin, Total Bilirubin, Direct Bilirubin, Indirect Bilirubin, Protein total, Albumin, Globulin, Alkaline Phosphatase, Glutamyl Transpeptidase, Urea Nitrogen, Creatinine, Cholesterol, Triglycerides, Glucose, Creatine Kinase, Creatine Phosphokinase MB Isoenzyme, Lactate Dehydrogenase, Calcium, Phosphorus, α -Amylase, Sodium, Potassium, Chloride, Albumin/globulin ratio.

<u>Urinalysis</u>: Appearance, Blood, Nitrite, Ketone, Protein, Glucose, Leukocytes, pH, Microscopic examination (Microscopic examination will be performed if dipstick test is positive for leukocytes, blood, nitrites, or proteins).

All hematology, biochemistry and urinalysis quantitative parameters will be summarized using descriptive statistics overall and by treatment sequence for each group at baseline and at end of study visit with raw data and change from baseline.

For all hematology and biochemistry parameters, frequency tables based on the classification of values as Low, Normal, High and Missing with respect to the reference ranges will be summarized by treatment sequence at baseline and end of study for each group. Frequency tables of urinalysis will be summarized by treatment sequence at baseline and end of study for each group, based on different types of classification rules. For urinalysis parameter, pH, the classification of values as

Low, Normal, High and Missing will be applied. For urinalysis parameters, Blood, Nitrite, Ketone, Protein and Glucose, the classification of values as Normal/-, +-, +, +++, ++++ will be applied. For urinalysis parameters, Appearance and Microscopic Examination, the classification of values as Normal, Abnormal, Missing, or Total will be applied. For urinalysis parameters, Leukocytes, the classification of values as Not Negative, Negative, Missing and Total will be applied.

In addition, shift tables from baseline to end of study for all hematology, biochemistry and urinalysis will be summarized and presented by treatment sequence for each group at End of Study.

All marked abnormal laboratory values will be listed by subject, treatment sequence and group.

All data will be listed by group, treatment sequence, subject, treatment, visit, and time point.

## 17.4 Vital Signs

The following Vital Signs measurements will be reported for this study:

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Pulse Rate (bpm)
- Temperature (<sup>0</sup>C)
- Respiratory Rate (breaths/min)

Systolic and diastolic blood pressures (mmHg) and pulse rate (beats/min) measurements as well as body temperature (°C) and respiration (breaths/min) will be presented by descriptive statistics overall and by treatment sequence for each group at baseline and end of study visit, and by group, treatment and time point for the values obtained during the treatment periods as raw data and change from baseline in the corresponding treatment period.

Frequency tables based on the classification of values as Low, Normal, High and Missing with respect to the reference ranges will be summarized by treatment sequence at end of study for each group, and by group, treatment and time point for the values obtained during the treatment period.

All marked abnormal for vital signs values will be listed.

All data will be listed by group, treatment sequence, subject, treatment, visit, and time point.

Markedly abnormal quantitative Vital Sign measurements will be identified in accordance with the following predefined markedly abnormal criteria:

| Variable | Unit | Low | High |
|------------------|------|----------------|-----------------|
| SBP | mmHg | < 85 mmHg | > 139 mmHg |
| DBP | mmHg | < 50 mmHg | > 90 mmHg |
| Pulse rate | bpm | < 50 Beats/min | > 100 Beats/min |
| Body temperature | °C | < 36 °C | > 37.3 °C |

## 17.5 Other Safety or Tolerability Evaluations

#### 17.5.1 ECG Evaluation

Results from the 12-Led Electrocardiogram (ECG) be presented by descriptive statistics overall and by treatment sequence for each group at baseline and end of study visit.

The following ECG parameters will be reported for this study:

- RR Interval (ms)
- PR Interval (ms)
- QRS Duration (ms)
- QT Interval (ms)
- QTc (Bazett) (ms)
- QTcF (Fridericia) (ms)
- Heart Rate (beats/min)
- Rhythm

Frequency tables for overall evaluation of ECG based on the classification of values as Normal, ANCS (Abnormal, Not Clinically Significant), ACS (Abnormal, Clinically Significant) and Missing will be presented by treatment sequence and overall for each group at the end of study visit.

12-lead ECG parameters and result of ECG will be listed in individual subject listing by group, treatment sequence, subject, visit, treatment and time point. All marked abnormal values of ECG evaluation will be listed by subject, treatment sequence and group.

# 17.5.2 Physical Examinations, and Chest X-ray

Full physical examination and chest X-ray examination will be performed, abnormal values will be marked in listing.

## 18 References

- 1. Valizadeh H, Nayyeri-Maleki P, Ghanbarzadeh S, et al. Pharmacokinetics and bioequivalence of two brands of metformin 500 mg tablets in Iranian healthy volunteers. J Pharmaceutical Investigation. 2014; 44(1):61-68.
- 2. Clinical Study Report EML056023-H105. "Randomized, open-label, 2-way, crossover, single oral-dose, fed, bioequivalence study between 500 mg Glucophage LCM 004 and 500 mg Glucophage® in healthy subjects". 2006.

# 1 Signature Page

Statistical Analysis Plan (29Jan2018, Final Version 1.0): MS200084\_0009

Shells (29Jan2018, Final Version 1.0): MS200084\_0009

A Randomized, Open-label, 2-way-crossover Study Assessing the Bioequivalence between Single Doses of 500 mg Glucophage Immediate Release (GIR) Tablets (Sino-American Shanghai Squibb Pharmaceuticals Ltd./ Manufactured in China) and 500 mg GIR Tablets (Merck Santé in Semoy/Manufactured in France) under Fed and Fasted State in Two Groups of Healthy Subjects

| PPD | |
|------------------------------|--------------------------|
| Trial Biostatistician | |
| Merck-Serono (Beijing) Pharm | naceutical R&D Co., Ltd. |
| Signature: | PPD<br>Date; .:x |
| PPD | |
| Trial Biostatistician | |
| PPD<br>Signature: | Date: PPD |
| PPD | |
| Senior Statistical Reviewer | |
| PPD<br>Siguature: | PPD<br>Date: . |
| CRO Pharmacokineticist | |
| PPD | |
| TU | |

PPD
CRO Biostatistician

PPD
PPD
PPD
PPD
Signature:
Date: ..